CLINICAL TRIAL: NCT02163265
Title: Impact of Surgical Treatments of Thoracic Deformation on Cardiopulmonary Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, Barbara Del Frari, MD, Associate Professor, Medical University Innsbruck
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20130111-621; KLI312 (Other Grant/Funding Number: FWF - Der Wissenschaftsfond)
Record Dates: First submitted 2014-03-21; First posted 2014-06-13 (Estimated); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Pectus Excavatum; Pectus Carinatum
MeSH Terms: conditions — Funnel Chest; Pectus Carinatum | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Surgery (Experimental): Patients suffering from Pectus excavatum and Pectus carinatum will be surgically treated
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Surgery — Patients suffering from Pectus excavatum Pectus carinatum will be treated surgically according to normal procedures

SUMMARY:
Pectus excavatum or carinatum are the most common congenital deformations of the ventral thoracic wall. Several different surgical methods with different techniques to correct these deformations have been described.

Some clinicians recommend a correction of the deformation to improve the cardiopulmonary efficiency. Other think that the correction has a more an aesthetic than a physiological benefit.

The aim of our prospective study is to evaluate whether patients with PE or PC are suffering preoperatively from a cardiopulmonary limitation at rest and under physical stress and if there is a change of cardiopulmonary function after the surgical correction.

DETAILED DESCRIPTION:
Pectus excavatum (PE) and pectus carinatum (PC) are the most common anterior chest wall deformities. Pectus excavatum, also known as funnel chest, is characterised by a deep depression usually involving the lower one-half to two-thirds of the sternum. PE is the most common congenital chest deformity and has a reported incidence of between 1:1000 and 8:1000 live births, with a male-to-female ratio of 3:1. Pectus carinatum, or pigeon breast, refers to protrusion of the sternum and is approximately seven times less frequent than PE, affecting 1:1000 to 1:10,000 live births. More than 26% have familial occurrence. The anatomic deformity is believed by many to be caused by a disproportionate growth of the costal cartilages as compared with the remainder of the bony thoracic skeleton, which exerts pressure on the sternum to cause depression (PE) and protrusion (PC). Although the majority of patients with PE are recognized during the first year of life, the depression usually becomes much more severe during childhood and adolescence; PC usually manifests itself at the time of a growth spurt in the early teenage years.

The deformities frequently present not only as an aesthetic disturbance, but also in association with mild limitation of activity, obstructive pulmonary mechanics, slight dyspnea, asthma, palpitations and abnormal cardiac physiology. Symptoms in PC patients remain often vague. PC patients usually complain more about the appearance of their chest rather than any functional difficulties. Chest wall deformities cause great social timidity, a sense of shame and often a feeling of limited self-worth and inferiority, depressive mood and inadequate social behaviour due to their disturbed body perception.

The results the investigators want to achieve with postoperative PFTs will demonstrate an improvement in total lung capacity and improved exercise performance and will show that both the restricted cardiac stroke volume and the increased work of breathing that have been described in PE patients can be ameliorated by operative intervention. These results will also contribute establish the criteria for the indication for surgery. The significant quality-of-life improvements perceived in psychosocial and physical functioning will encourage physicians to approach PE repair in the same manner as physicians do treatment of other deformities that have a deleterious impact on the psychological and physical well-being of the individual. Systematic evaluation of body image should become a diagnostic standard in the assessment of patients presenting themselves for correction of thoracic wall deformities.

ELIGIBILITY:
Inclusion Criteria:

* both women and men aged between 10 and 50 suffering from Pectus excavatum or Pectus carinatum

Exclusion Criteria:

* patients suffering from Poland Syndrome
* patients who already had a surgical PE corrections
* other surgical treatments of the thorax
* congenital heart defect
* existing contra-indication for anaesthesia
* body height less than 130 cm

Ages: 10 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2014-07; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Improvement of lung function from baseline | 6 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Del Frari, MD, Principal Investigator — Medical University Innsbruck
Locations (1):
- Medical University Innsbruck, Innsbruck, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Del Frari B, Blank C, Sigl S, Schwabegger AH, Gassner E, Morawetz D, Schobersberger W. The questionable benefit of pectus excavatum repair on cardiopulmonary function: a prospective study. Eur J Cardiothorac Surg. 2021 Dec 27;61(1):75-82. doi: 10.1093/ejcts/ezab296. PMID 34263302
- [Derived] Del Frari B, Sigl S, Schwabegger AH, Blank C, Morawetz D, Gassner E, Schobersberger W. Impact of surgical treatment of pectus carinatum on cardiopulmonary function: a prospective study. Eur J Cardiothorac Surg. 2021 Jan 29;59(2):382-388. doi: 10.1093/ejcts/ezaa335. PMID 33212487
- [Derived] Sigl S, Del Frari B, Harasser C, Schwabegger AH. The effect on cardiopulmonary function after thoracoplasty in pectus carinatum: a systematic literature review. Interact Cardiovasc Thorac Surg. 2018 Mar 1;26(3):474-479. doi: 10.1093/icvts/ivx353. PMID 29092017